CLINICAL TRIAL: NCT01979185
Title: A Phase 1, Randomized, Open-label, Cross-over Study to Evaluate the Pharmacokinetic Interaction Between SSP-004184 (SPD602) and Simvastatin in Healthy Adult Subjects
Brief Title: Effect of SSP-004184 (SPD602) on the Pharmacokinetics of Simvastatin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPD602-114
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Results first posted 2014-12-24 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Healthy
MeSH Terms: interventions — Simvastatin

ARMS (2):
- Simvastatin (Active Comparator): Administered as a single oral 20 mg dose on Day 1.
  Interventions: Drug: Simvastatin
- Simvastatin + SSP-004184SS (Experimental): Simvastatin (20 mg) + SSP-004184SS (30 mg/kg) administered concomitantly as a single oral dose on Day 1.
  Interventions: Drug: Simvastatin; Drug: SSP-004184SS

INTERVENTIONS:
Drug: Simvastatin
Drug: SSP-004184SS
  Other Names: SPD602
  Arms: Simvastatin + SSP-004184SS

SUMMARY:
This is a randomized, open-label study to evaluate the effect of a single dose of SSP-004184 on the pharmacokinetics of a single dose of simvastatin in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy male and female volunteers
* Serum ferritin, hemoglobin and erythrocyte indices within normal range

Exclusion Criteria:

* Evidence of any active or chronic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2013-12-13 (Actual); Study Completion 2013-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Clinical Pharmacology of Miami, Inc., Miami, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin First: Subjects received Simvastatin 20mg in Period 1, followed by Simvastatin 20mg and SSP-004184SS 30mg/kg during Period 2.
- Simvastatin + SSP-004184SS First: Subjects received Simvastatin 20mg and SSP-004184SS 30mg/kg in Period 1, followed by Simvastatin 20mg during Period 2.
Period: Period 1
Arm/Group | Simvastatin First | Simvastatin + SSP-004184SS First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Simvastatin First | Simvastatin + SSP-004184SS First
Started | 15 | 15
Completed | 15 | 14 (1 subject discontinued due to a positive drug test prior to receiving Simvastatin alone in Period 2.)
Not Completed | 0 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set: All subjects who had taken at least 1 dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin First | Simvastatin + SSP-004184SS First | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.1 (14.97) | 39.6 (15.9) | 39.3 (15.17)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 6 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) for Simvastatin
Description: AUCinf is the area under the plasma concentration versus time curve extrapolated from time 0 to infinity, calculated using the observed value of the last nonzero concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: Study Periods 1 & 2: Within 30 minutes pre-dose, and Post-dose 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72 hours.
Population: Pharmacokinetic Set: All subjects who took at least 1 dose of investigational product and for whom the primary pharmacokinetic data were considered sufficient and interpretable.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- Simvastatin Alone: Administered as a single oral 20 mg dose on Day 1.
Arm/Group | Simvastatin Alone | Simvastatin + SSP-004184SS
Number analyzed (Participants) | 27 | 29
ng*h/ml | 38.142 (19.239) | 26.601 (17.864)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Simvastatin + SSP-004184SS; The means of the log-transformed pharmacokinetic parameters were compared between treatments using a mixed-effects model with period and treatment as fixed effects, and subject nested within sequence as a random effect. In order to estimate the magnitude of the treatment regimen differences in pharmacokinetic parameters, the geometric mean ratio (i.e., the least squares mean difference in the log-transformed parameters back transformed to the original scale) and their 90% CIs were calculated; Test type: Non-Inferiority or Equivalence — If the 90% CI of the geometric mean ratios fell within the range (0.80, 1.25), then equivalence was assumed and the hypothesis that a drug interaction occurred was rejected. If the 90% CIs were not wholly contained within the range (0.80, 1.25), then a drug interaction was not excluded; Mixed-effects Model; Ratio of Geometric LS Means = 0.632, 90% CI 2-sided [0.538 to 0.744]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Measureable Concentration (AUClast) of Simvastatin
Description: AUClast is the area under the concentration versus time curve from the time of dosing to the last measurable concentration. AUC can be used as a measure of drug exposure. It is derived from drug concentration and time so it gives a measure how much and how long a drug stays in a body.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | Simvastatin Alone | Simvastatin + SSP-004184SS
Number analyzed (Participants) | 29 | 30
ng*h/ml | 34.351 (18.911) | 24.019 (16.701)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Simvastatin + SSP-004184SS; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed-effects Model; Ratio of Geometric LS Means = 0.630, 90% CI 2-sided [0.543 to 0.730]

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Simvastatin
Description: Cmax is a term that refers to the maximum (or peak) concentration that a drug achieves in the body after the drug has been administrated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Simvastatin Alone | Simvastatin + SSP-004184SS
Number analyzed (Participants) | 29 | 30
ng/mL | 5.006 (3.125) | 2.72 (1.265)
Statistical Analysis 1: Comparison: Simvastatin Alone vs Simvastatin + SSP-004184SS; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Mixed-effects Model; Ratio of Geometric LS Means = 0.594, 90% CI 2-sided [0.526 to 0.672]

ADVERSE EVENTS:
Arm/Group | Simvastatin Alone | Simvastatin + SSP-004184SS
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 1/29 | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin Alone (N=29) | Simvastatin + SSP-004184SS (N=30)
Headache (Nervous system disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.